CLINICAL TRIAL: NCT02315170
Title: Assessment of Novel Intraocular Injection Guide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maturi, Raj K., M.D., P.C. (Individual)
Responsible Party: Principal Investigator, Raj Maturi, President, Maturi, Raj K., M.D., P.C.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: rkm006
Record Dates: First submitted 2014-12-09; First posted 2014-12-11 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-05

CONDITIONS: Retinal Disease
Keywords: diabetic retinopathy; age-related macular edema
MeSH Terms: conditions — Retinal Diseases; Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intraocular injection guide (Experimental): novel intraocular injection guide is a long, tubular structure consisting of a non-moldable material with a single internal opening. There is a 2x2 square hole located at the bottom of the device where the needle exits the guide and enters the eye
  Interventions: Device: intraocular injection guide
- standard lid speculum (Active Comparator): Standard wire eyelid speculum
  Interventions: Device: standard lid speculum

INTERVENTIONS:
Device: intraocular injection guide — The device is 35mm long with tapered edges for an easy grip and it aligns with the curvature of the cornea to ensure that needle entry takes place at the optimal distance for injection
  Arms: intraocular injection guide
Device: standard lid speculum — standard wire lid speculum
  Arms: standard lid speculum

SUMMARY:
To determine if a novel intraocular injection guide (IIG) reduces patient discomfort during and after intravitreal injections.

DETAILED DESCRIPTION:
This study is being conducted to assess the potential for an intraocular injection guide to increase comfort levels both during and after such injections. The hypothesis is that patients will feel increased comfort from a device which eliminates the need for a speculum while still keeping the eyelids apart, allowing a physician to deliver treatment. The results of this study will allow physicians to select the optimal device for patient comfort and well-being during intravitreal injections

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be receiving bilateral injections of the same dose of vascular endothelial growth factor (VEGF) inhibitor
* Injections in both eyes must be given on the same day
* Male or female age 18 years or older

Exclusion Criteria:

-Any condition or reason that precludes the subject's ability to comply with the study -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj K Maturi, MD, Principal Investigator — Raj K. Maturi, MD, PC
Locations (1):
- Raj K Maturi MD PC, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: all subjects presenting for bilateral injection were offered the chance to participate in this clinical trail
Pre-assignment Details: eyes were chosen for the novel guide or standard lid speculum using a randomizing table
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Intraocular Injection Guide | Standard Lid Speculum
Started (Each participant will have one eye randomly selected to receive Intraocular Injection Guide and the other eye will receive Standard Speculum.) | 50; 50 eyes | 50; 50 eyes
Completed | 50; 50 eyes | 50; 50 eyes
Not Completed | 0; 0 eyes | 0; 0 eyes

BASELINE CHARACTERISTICS:
Population: Only subjects needing bilateral ocular injections were included in the study.The total number of participants was 50 (100 eyes). Baseline characteristics were identical in both groups.One eye received the treatment with the injection guide while the fellow eye received the treatment with a standard lid speculum.
Groups:
- All Participants: Only subjects needing bilateral ocular injections were included in the study. The total number of participants was 50 (100 eyes). Baseline characteristics were identical in both groups. One eye received the treatment with the injection guide while the fellow eye received the treatment with a standard lid speculum.
Arm/Group | All Participants
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 30
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 15

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS)
Description: The VAS is a horizontal line, 100 mm in length, and anchored by word descriptors at each end. The scale scores range from 0mm (no pain) to 100mm (very severe pain). The patient marks on the line the point that they feel represents their perception of their current state (no pain to very severe pain).
Time Frame: one time for about 30 sec or less
Population: Total number of subjects is 50 - however as the system here is designed for whole body count (not bilateral organs such as eyes), the total number will appear to be double of actual number of subjects.
Measure: Median (Standard Deviation); unit: mm on the VAS
Units Other Than Participants: eyes
Arm/Group | Intraocular Injection Guide | Standard Lid Speculum
Number analyzed (Participants) | 50 | 50
Number analyzed (eyes) | 50 | 50
mm on the VAS | 14 (6) | 33 (7)

ADVERSE EVENTS:
Arm/Group | Intraocular Injection Guide | Standard Lid Speculum
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
This is a small one event study (about 10 min duration). The participant evaluates which speculum (used for about 30 sec or less) during the procedure provides better comfort. Thus, long term evaluation has not been peformed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes